CLINICAL TRIAL: NCT03654092
Title: Effects of a Long-term Home-based Exercise Training Program Using Minimal Equipment vs Usual Care in COPD Patients: A Multicenter Randomized Controlled Trial
Brief Title: Home-based Exercise Training for COPD Patients (HOMEX-2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HOMEX-2
Record Dates: First submitted 2018-07-17; First posted 2018-08-31 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Chronic Disease; Lung Diseases, Obstructive; Respiratory Disease
Keywords: Exercise; Minimal equipment; Home-based; COPD; Exercise training intervention; Randomized controlled trial
MeSH Terms: conditions — Chronic Disease; Lung Diseases, Obstructive; Respiration Disorders; Motor Activity; Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): Home-based, minimal equipment exercise training program.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Usual care (study participation does not have any impact on regular treatment decisions, including participation in other exercise training programs).

INTERVENTIONS:
Behavioral: Exercise — Home-based exercise training program that requires only minimal equipment, and is individually adaptable to the participant's exercise level (6 times per week; 15-20 min; 38 exercise cards and one interactive training agenda booklet). After randomization, a health care professional (HOMEX coach) will visit the intervention group participants at their home to set up the training location, to instruct the exercises and to establish individualized goals. Follow-up visits are planned after 3 and 8-9 weeks. Regular telephone calls will be conducted by the same HOMEX coach to motivate the patients, to discuss training progress and concrete benefits and barriers, and to adapt goals and the training program. Additional intervention elements are that a relative or friend is involved as a "sparring" partner to support the participant. The general practitioner is informed about the participation of his/her patient in the intervention.
  Arms: Exercise intervention

SUMMARY:
The aim of this study is to assess the effectiveness of a home-based exercise training program in COPD patients who did not participate in an inpatient or outpatient rehabilitation program within the last 2 years.

DETAILED DESCRIPTION:
Exercise training is an important component of pulmonary rehabilitation (PR) the management of chronic obstructive pulmonary disease (COPD) and numerous trials have shown large improvements in health-related quality of life (HRQoL) and exercise capacity in persons with COPD. However, the great majority of patients who would benefit from PR never follow such a program. Moreover, many COPD patients are either not instructed to exercise at all or fail to adhere to exercise training at home after completing PR.

This study evaluates a newly developed exercise training program that requires minimal equipment (i.e., only a chair and elastic bands) and can be easily implemented long-term in the patient's home-setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent after being informed
* Diagnosis of COPD, defined as forced expiratory volume in 1s/forced vital capacity (FEV1/FVC)<70% predicted, FEV1<80 % predicted after bronchodilation, with or without chronic symptoms (cough, sputum production) corresponding to a GOLD stage II-IV
* No participation in an inpatient or outpatient pulmonary rehabilitation within the last 12 months
* Male and female patients ≥40 years of age
* Knowledge of German language to understand study material and assessments

Exclusion Criteria:

* Patients not able to conduct the exercise training program due to physical, cognitive or safety reasons, as judged by investigator; e.g., lower limb joint surgery within preceding 3 months, unstable cardiac disease, predominant neurological limitations.
* Planned participation in a pulmonary rehabilitation program

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea (Chronic Respiratory Questionnaire (CRQ) domain) | Change from baseline to 12 months
  Dyspnea domain of the CRQ; 5 questions; 7-point Likert-type scale ranging from 1 (most severe dyspnea) to 7 (no dyspnea)

SECONDARY OUTCOMES:
Dyspnea (Chronic Respiratory Questionnaire (CRQ) domain) | Change from baseline to 3, 6 and 12 months
  Dyspnea domain of the CRQ; 5 questions; 7-point Likert-type scale ranging from 1 (most severe dyspnea) to 7 (no dyspnea)
Functional exercise capacity (Six-Minute Walk Test; 6MWT) | Change from baseline to 12 months
  Total distance in meters walked by the patient during timed six minutes. The 6MWT will be conducted twice (the better result will be used) and according to the American Thoracic Society (ATS) guidelines
Functional exercise capacity (1-min Sit-to-Stand test; 1-min-STS test) | Change from baseline to 12 months
  The number of repetitions that the patient completes the full sit-to-stand movement from a standard chair (i.e. standing up from a chair and sitting down again) during one minute
Health-related quality of life (Chronic Respiratory Questionnaire; CRQ) | Change from baseline to 12 months
  Remaining domains of the CRQ (besides the dyspnea domain): Domains fatigue, emotional function and mastery. The total CRQ contains 20 questions responded to on a 7-point Likert-type scale, ranging from 1 to 7 with lower scores indicating worse HRQoL, loading on the domains dyspnea, fatigue, emotional and mastery
Physical activity (PROactive physical activity in COPD instrument, clinical visit version; C-PPAC; domains amount and difficulty) | Change from baseline to 12 months, measured during 1 week prior to the visits
  The C-PPAC is a validated and reliable hybrid tool combining a short patient-reported outcome questionnaire and two activity monitor variables (assessed by the accelerometer ActiGraph®) to measure physical activity in COPD patients in the two domains amount and difficulty (item scores 0-4, scale 0-100)
Symptoms (COPD Assessment Test; CAT) | Change from baseline to 12 months
  The CAT measures the impact of COPD on a person's health status (8 questions, 6-point Likert-type scale)
Hospital Anxiety and Depression Scale (HADS) | Change from baseline to 12 months
  Symptoms of depression and anxiety (14 questions, 4-point Likert-type scale)
Health status (Feeling Thermometer; FT) | Change from baseline to 12 months
  The FT is a visual analogue scale for overall health state ranging from 0 (worst health you can imagine) to 100 (best healthy you can imagine)
Health-related quality of life (EuroQOL; EQ-5D-5L) | Change from baseline to 12 months
  The EQ-5D-5L assesses the 5 dimensions mobility, self-care, usual activities, pain/discomfort, anxiety/depression including 1 item with 5 levels each
Exacerbations of COPD (event based, patient reported) | During the entire study, assessed at 3, 6 and 12 months
  The event-based definition required an increase in symptoms and an increase in dosage of or new prescription of systemic corticosteroids and/or antibiotics

OTHER OUTCOMES:
Compliance to the exercise training program | Assessed daily by intervention group participants during 12 months
  Percentage of fulfilled training sessions based on training diaries
Satisfaction with the exercise training program (self-developed questionnaire) | From baseline to 12 months, assessed at 12 months
  Self-developed questionnaire assessing satisfaction with the intervention: 10 specific questions regarding elements of the intervention using Likert-type scales from 0=not useful at all to 10=very useful) and 4 global questions using Likert-type scales (from 0=worst outcome to 4=best outcome)
Experience with the exercise training program of the participants | From baseline to 12 months, assessed at 12 months
  Semi-structured interview and/or focus groups
Experience with the exercise training program of the health professionals | From baseline to 12 months, assessed at 12 months
  Semi-structured interview and/or focus groups
Cost effectiveness | From baseline to 12 months, assessed at 3, 6 and 12 months
  Questionnaire: Cost per quality-adjusted life-year, direct healthcare costs, direct non-healthcare costs, indirect costs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Frei A, Radtke T, Dalla Lana K, Braun J, Muller RM, Puhan MA. Effects of a long-term home-based exercise training programme using minimal equipment vs. usual care in COPD patients: a study protocol for two multicentre randomised controlled trials (HOMEX-1 and HOMEX-2 trials). BMC Pulm Med. 2019 Mar 1;19(1):57. doi: 10.1186/s12890-019-0817-7. PMID 30823913